CLINICAL TRIAL: NCT06416033
Title: Serum Irisin Level In Leprosy Patients
Status: Completed | Type: Observational
Sponsor: Aswan University (Other)
Responsible Party: Principal Investigator, Esraa Nagy Zaki Faheem, Resident at Dermatology, Venereology and Andrology, Aswan University
Other Study IDs: Irisin Level In Leprosy
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-05

CONDITIONS: Leprosy
Keywords: Leprosy; Irisin; tuberculoid leprosy; lepromatous leprosy
MeSH Terms: conditions — Leprosy; Leprosy, Tuberculoid; Leprosy, Lepromatous

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A :(Leprosy Group): About 29 patients newly affected with Leprosy and The plasma irisin level of the participants will be measured by enzyme-linked immunosorbent assay (ELISA).
  Interventions: Procedure: Serum Irisin
- Group B:(Control Group): About 29 apparently healthy individuals and The plasma irisin level of the participants will be measured by enzyme-linked immunosorbent assay (ELISA).
  Interventions: Procedure: Serum Irisin

INTERVENTIONS:
Procedure: Serum Irisin — Measurement of plasma irisin level in leprosy patients.

SUMMARY:
* Measurement of plasma irisin level in leprosy patients.
* Correlation of plasma irisin level between leprosy patients and healthy controls.
* Correlation of plasma irisin level in different leprosy types.

DETAILED DESCRIPTION:
Leprosy is a chronic granulomatous infectious disease which infects mainly superficial peripheral nerves, mucosa of upper respiratory tract, testicles, bones, and eyes. It's an intracellular infection caused by the acid-fast bacillus, Mycobacterium leprae.

Both age and sex are important risk factors for leprosy infection, adolescents aged between 10 and 19 years and adults aged more than 30 years are more liable to leprosy, and the possibility of leprosy infection of adult males is twice as much as adult females.

Leprosy evolution involves complex host immune mechanisms that influence the clinical presentation of the disease . the spectral pathology of leprosy can be diagnosed by using two coexisting classification systems. The WHO classification system which is based on the number of lesions and Ridley and Jopling classification system which is based on the histopathology .

The WHO classification system includes individuals with more than five lesions which are classified as multibacillary (MB) patients, and individuals with less than five lesions which are classified as paucibacillary (PB) patients .While Ridley and Jopling classification system includes tuberculoid leprosy (TT), lepromatous leprosy (LL) and borderline phenotypes: {borderline tuberculoid (BT), mid-borderline (BB), and borderline lepromatous (BL).

Tuberculoid leprosy (TT) is characterized by the presence of one to three cutaneous lesions, called plaques. These lesions are circular or oval, erythematous/hypopigmented, hairless, scaly, dry and anesthetic. On the other hand, lepromatous leprosy (LL) is characterized by extensive and multiple bilateral lesions, which may include macules, papules, nodules, and plaques .

The majority of patients, however, present with the borderline phenotypes. In these phenotypes, the bacterial load correlates with the histological features, borderline tuberculoid (BT) being more closely related to tuberculoid leprosy( TT) patients while borderline lepromatous (BL) to lepromatous leprosy (LL) patients. The borderline states are immunologically unstable and susceptible to the occurrence of leprosy reactions.

In 1991 the World Health Assembly decided to 'eliminate leprosy as a public health problem' by the year 2000. Elimination was defined as decreasing the disease prevalence globally to less than 1 case per 10,000 populations. In 2000 the World Health Organization (WHO) announced that elimination was reached globally.

Irisin is a protein formed of 112 amino acids. It was discovered in 2012 at Harvard University. And named after an ancient Goddess called Iris, who served as a messenger among the Gods in Greek mythology.

Irisin has been linked to many metabolic diseases, including obesity, lipid metabolism ,cardiovascular disease (CVD), type 2 diabetes mellitus (T2DM) ,polycystic ovary syndrome (PCOS) ,Nonalcoholic fatty liver disease (NAFLD) and metabolic bone diseases .

ELIGIBILITY:
Inclusion Criteria:

- New cases of leprosy patients.

Exclusion Criteria:

* Old cases with leprosy.
* Patients with cardiovascular disease (CVD) and type 2 diabetes mellitus (T2DM).
* Patients with polycystic ovary syndrome (PCOS), Nonalcoholic fatty liver disease (NAFLD) and metabolic bone diseases.

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study will include patients with leprosy and healthy controls attending in the outpatient clinic of Dermatology, Venereology and Andrology, Aswan University Hospital, Aswan University.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
measurement of Serum Irisin | 24 hours
  comparing the plasma irisin levels in leprosy patients with healthy Participants

CONTACTS AND LOCATIONS:
Overall Officials: Moustafa El Taieb, Professor, Study Chair — Department of Dermatology, Venereology and Andrology Faculty of Medicine, Aswan University
Locations (1):
- Aswan University Hospital, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: Undecided